CLINICAL TRIAL: NCT05806151
Title: Oligo-metastatic neoPlasms From the gastRo-intEstinal Tract: iDentIfiCaTIon Of cliNical and Molecular Drivers: the PREDICTION Study
Brief Title: Prediction of True Oligo-metastatic Disease.
Acronym: PREDICTION
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: NCINaples
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Oligometastatic Disease
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — FFPE tissues.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Genetic and immunologic assessments — Definitive Local Therapies including surgery, radiotherapy, radio-frequency ablation of metastases.

SUMMARY:
In recent years, the scientific community has recognized the need to differentiate between poly- and oligo-metastatic disease (OMD) in oncology due to their distinct clinical and biological behavior. The definition of "true" and good-prognosis OMD is necessarily retrospective, as many patients initially considered oligo-metastatic develop poly-metastatic disease within one year. The PREDICTION study is a prospective, observational, and monocentric investigation. The study has two primary objectives. The first one is descriptive and aims to determine the prevalence of specific biological characteristics in OMD derived from gastrointestinal tract neoplasms (colon, stomach, biliary tract, exocrine glands of the digestive tract). These biological characteristics include genetic landscape and T lymphocyte infiltrate of the primary tumor and/or metastases. Genetic assessment will be done on formalin-fixed paraffin-embedded (FFPE) tissues or liquid biopsies with the Oncomine Solid Tumour DNA kit (Thermo Fisher Scientific, Waltham, MA, USA). Data analysis will be performed using the Torrent Suite Software v5.0 (Thermo Fisher Scientific). The analysis of T lymphocytes will be conducted through immunohistochemistry (IHC) in primary and or metastatic tissues (if available). The second co-primary objective aims to identify OMD through the prognostic effect of a score designed ad hoc. It is tested in a single pathology, namely in patients with metastatic colorectal cancer. A score is constructed based on the following characteristics, with possession of all characteristics (3+) constituting the full score: a primitive/metastasis genetic concordance >80% = 1 point; high T-lymphocyte infiltration GRZB+ (>10 cells/mm2) in the primary tumor and/or metastases (where tissue is available) = 1 point; absence of clonal evolution favoring specific key-driver genes = 1 point. The hypothesis is that patients with true OMD (score 3+) have a significantly lower rate of progression at one year, defined as recurrence after radical surgery or progression (in oligometastatic patients who are not candidates for upfront definitive local treatment) based on RECIST v 1.1 criteria since enrollment in the study, compared to those with false OMD who subsequently develop polymetastatic disease. The treatments will be chosen at the discretion of the referring Oncologist, in multidisciplinary sessions, according to normal clinical practice. The sample size was determined using a two-sided test of difference between proportions to evaluate the statistical significance of the difference in recurrence within 1 year. For this purpose, the following scenario was considered: a reasonable probability of the simultaneous occurrence of the 3 factors in true OMD (score 3+) of 60%; a recurrence rate of 20% for true OMD (score 3+), and 80% for false OMD (score <3+). With a significance level of α=0.05, a test power of 90%, and a Fisher exact test, the required number of patients to be enrolled is 32, to be recruited over an expected period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study must meet the following criteria:
* Diagnosis of gastroenteric tumors (colon, stomach, biliary tract, exocrine glands of the digestive tract);
* OMD: one to three lesions per organ with a maximum tumor diameter of less than 70 mm and no lesion with a diameter greater than 25 mm;
* Availability of FFPE (Formalin Fixed Paraffin Embedded) inclusions from resected primary tumor;
* Written informed consent.

Exclusion Criteria:

* Previous or concurrent malignant neoplasms;
* Presence of cerebral metastases;
* Refusal or inability to provide informed consent;
* Inability to guarantee follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients affected by gastroenteric tumors (colon, stomach, biliary tract, exocrine glands of the digestive tract) with oligo-metastatic disease. Oligometastatic patients will be defined as those presenting with one to three lesions per organ with a maximum tumor diameter of less than 70 mm and no lesion with a diameter greater than 25 mm.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Progression/Recurrence | 1 year
  Rate of recurrence/progression within one year

CONTACTS AND LOCATIONS:
Locations (1):
- Alessandro Ottaiano, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ottaiano A, De Luca A, Santorsola M, Scognamiglio G, Di Mauro A, Chiodini P, Lambiase M, Sacco A, Petrillo A, Granata V, Fusco R, Mercadante E, Martucci N, De Luca G, Rocca A, Celentano E, Crispo A, Di Gennaro P, Tatangelo F, Ferrara G, Izzo F, Belli A, Patrone R, Delrio P, Rega D, De Franciscis S, Muto P, Ravo V, Di Franco R, Borzillo V, Santagata S, Rea G, Castaldo D, Pace U, De Feo G, Scala S, Nasti G, Normanno N. Oligo-metastatic neoPlasms from the gastro-intestinal tract: iDentIfiCaTIon of cliNical and molecular drivers: the PREDICTION study. BMC Cancer. 2023 Oct 19;23(1):1010. doi: 10.1186/s12885-023-11479-w. PMID 37858132